CLINICAL TRIAL: NCT06647680
Title: Neoadjuvant Chemotherapy and Tislelizumab (PD-1 Inhibitior) for Locally Advanced Rectal Cancer: a Single-center, Prospective, Phase II Study
Brief Title: Neoadjuvant Chemotherapy and PD-1 Inhibitor for Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QYFYEC2024-181
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-09

CONDITIONS: Rectal Cancer Patients
Keywords: Rectal cancer; Chemotherapy; Tislelizumab; Complete response; Recurrence free survival
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response | interventions — Chemoradiotherapy; Oxaliplatin; Capecitabine; Immune Checkpoint Inhibitors; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with rectal cancer receiving neoadjuvant chemotherapy and PD-1 inhibitor (Experimental): Experimental: Combination of drugs prior to surgery Receive the experimental combination of drugs (chemoradiation (Oxaliplatin and Capecitabine) + PD-1 inhibitor (Tislelizumab) for 3 cycles prior to surgery and undergo laboratory tests and study procedures on specified days during the study period, complete end of study evaluations and tests, and participate in post-study follow up every three months for three to four years. The time in the study will take approximately four - six hours during pre-study, study and end of study visits.
  Interventions: Drug: Receive the experimental combination of drugs (chemoradiation (Oxaliplatin and Capecitabine) + PD-1 inhibitor (Tislelizumab) for 3 cycles

INTERVENTIONS:
Drug: Receive the experimental combination of drugs (chemoradiation (Oxaliplatin and Capecitabine) + PD-1 inhibitor (Tislelizumab) for 3 cycles — Receive the experimental combination of drugs (chemoradiation (Oxaliplatin and Capecitabine) + PD-1 inhibitor (Tislelizumab) for 3 cycles prior to surgery and undergo laboratory tests and study procedures on specified days during the study period, complete end of study evaluations and tests, and participate in post-study follow up every three months for three to four years. The time in the study will take approximately four - six hours during pre-study, study and end of study visits.

SUMMARY:
To evaluate the safety and preliminary efficacy of preoperative chemotherapy and PD-1 inhibitor Tislelizumab for Rectal Cancer patients.Go through laboratory and medical tests to verify eligibility to enter the study, receive the experimental combination of drugs CAPOX (Oxaliplatin and Capecitabine) for 3 cycles prior to surgery and undergo laboratory tests and study procedures on specified days during the study period, complete end of study evaluations and tests, and participate in post-study follow up every three months for three years.

DETAILED DESCRIPTION:
Treatment will continue until participants experiences disease progression, unacceptable toxicity or withdraws consent and will include chemotherapy and PD-1 inhibitor (Tislelizumab) x 3 cycles (9 weeks). For participants experiencing unacceptable CAPOX or Tislelizumab related toxicity, yet obtaining therapeutic benefit, participants will be allowed to continue treatment, if well tolerated at the discretion of the investigator.After the completion of 3 cycles of treatment, the patients will rest for 2 weeks and then undergo surgery, and adjuvant therapy will be decided according to the postoperative pathology.

Upon discontinuation of study treatment, participants will receive safety follow-up assessments approximately 30 and 90 days later. Once the 90-day safety follow-up is complete, participants will enter the survival follow-up period where they will continue to be followed approximately every three months until death, withdrawal of consent, or overall study completion. Patients will be followed for survival for 36 months from enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial
* Age 18 years or greater
* Pathologically proven diagnosis of adenocarcinoma of the rectum
* Clinically determined to be stage T3 or T4, N0-N2, and M0
* Be fully active, able to carry on all pre-disease performance without restriction or Restricted in physically strenuous activity.
* Contrast-enhanced imaging of the abdomen and chest by CT to exclude distant metastases and provide local tumor stage
* Preoperative ECOG status score 0-1
* Preoperative ASA grade I-III
* Adequate bone marrow function
* Adequate renal and liver function
* No active second cancers
* Be willing and able to comply with all aspects of the protocol
* Women of childbearing potential must have used reliable contraception or have had a pregnancy test result within 7 days prior to enrollment. Be negative and willing to use an adequate method of contraception for the duration of the trial and for 8 weeks after the last administration of the trial drug.
* Adequate bone marrow function defined as follows: Absolute neutrophil count (ANC) ≥ 1,200 cells/mm3 Platelets ≥ 100,000 cells/mm3 Hemoglobin ≥ 8.0 g/dl.
* Adequate hepatic function within within 28 days before registration on this study:total bilirubin must be ≤ ULN (upper limit of normal) for the lab unless the patient has a bilirubin elevation > ULN to 1.5 x ULN due to Gilbert's disease or similar syndrome involving slow conjugation of bilirubin; and AST and ALT must be ≤3 x ULN for the lab If AST and/or ALT is ≥ ULN but ≤ 3 x ULN, serologic testing for Hepatitis B and C must be performed and results for viral infection must be negative.
* Adequate renal function within 28 days before randomization defined as serum creatinine ≤ 1.5 x ULN for the lab or calculated creatinine clearance > 30 mL/min

Exclusion Criteria:

* Age less than 18 years
* Pregnant or breastfeeding women
* Prior invasive malignancy unless disease free for a minimum of three years
* Preoperative body temperature ≥ 38°C or concurrent infectious diseases requiring systemic therapy;
* Severe mental illness;
* Severe abnormal heart, lung and kidney function
* History of unstable angina pectoris or myocardial infarction within 6 months;
* History of cerebral infarction or cerebral hemorrhage within 6 months;
* Patients with abnormal coagulation function;
* Have a history of psychotropic drug abuse or have a mental disorder;
* Continuous use of glucocorticoids within 1 month (except topical application);
* Patient has participated in or is participating in other clinical studies (within 6 months);
* According to the judgment of the investigator, it endangers the patient's health or affects the experimental results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response and pathological complete response | The cCR was evaluated at 8 weeks after neoadjuvant chemotherapy. The pCR was evaluated after surgery.
  The cCR is judged by imaging (CT/MRI), tumor markers, and colonoscopy. The pCR is examined by pathological examination.

IPD SHARING:
Plan to Share IPD: No